CLINICAL TRIAL: NCT00348621
Title: Clinical Trial of Interventions for Visual Loss in Nursing Home Residents
Brief Title: A Study of Interventions to Reduce Disability From Visual Loss in Nursing Home Residents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AG015812 (NIH); R01AG015812 (NIH)
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Cataract; Refractive Error; Low Vision
Keywords: cataract surgery; refractive correction; low vision services; nursing home; visual impairment
MeSH Terms: conditions — Cataract; Refractive Errors; Vision, Low; Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Visual impairment intervention program (Active Comparator): enhanced access to eye care services
  Interventions: Procedure: Visual impairment intervention program
- Usual care (No Intervention): family and nursing home was apprised of ocular exam results; eye care services left to family/nursing home arrangements

INTERVENTIONS:
Procedure: Visual impairment intervention program — enhanced access to eye care services
  Arms: Visual impairment intervention program

SUMMARY:
The purpose of this clinical trial is to determine if interventions within the nursing home to restore vision, or cope with visual loss, in residents with visual impairment result in improvement or less decline in mobility scores, and socialization scores, compared to residents with visual impairment in nursing homes with no such intervention. The investigators hypothesized that nursing home residents with visual loss who receive cataract surgery, or refractive correction, or low vision aids would have have better socialization scores and mobility scores at 6 months and 12 months compared to nursing home residents with visual impairment who are advised to seek services, but have no specific program.

DETAILED DESCRIPTION:
The goal of this project was to quantify the impact of visual acuity impairment on socialization and physical function of nursing home residents, and to determine the cost effectiveness of a visual impairment intervention program designed to enhance access to eye care services. To accomplish these aims, the investigators enrolled a complete sample of visually impaired persons from 28 nursing homes in the Lower Eastern Shore of Maryland and Delaware. From the same facilities, the investigators also enrolled a random sample of non-visually impaired residents, with sample size equal to the sample of visually impaired. The group of visually impaired residents was randomized (by facility) to an intervention program or "usual care" group. The intervention program facilitated the utilization of eye care services of the three main causes of visual impairment: refractive error, cataract, and low vision associated with age-related eye diseases. All study groups provided data at baseline, six and twelve months from intervention, and data on eye care utilization, hospitalizations, use of psychoactive medications and mortality collected every other month (bi-monthly). Patients had a screening test of visual acuity, using standard letter/symbol charts, and grating charts. The mental status was tested using the MiniMental State Examination. Social function, physical function, and mobility were assessed through questionnaires asked of nursing home staff familiar with the patient, and the questions were modeled on the Minimum Data Set questions or specially designed for nursing home residents.

The investigators compare the mobility scores, and socialization scores, of nursing home residents with visual loss randomized to the intervention homes to the scores of nursing home residents with visual loss randomized to control homes. The investigators use the mobility and socialization scores of those without visual loss at baseline and follow up to compare with the trajectory of decline in those with visual loss.

ELIGIBILITY:
Inclusion Criteria:

* Nursing homes in Eastern Shore of Maryland,within 1.5 hour drive of Salisbury MD
* Nursing home administrators and resident committees approved the study
* Nursing home residents:
* Age 65 and older
* more than 30 day length of Stay
* Capable of acuity testing

Exclusion Criteria:

* Nursing home residents:
* staff assessment noted imminent death likely (within 3 months)
* resident unable to provide informed consent and guardian not locatable
* resident's only language was not understood by nursing staff

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2544 (Actual)
Dates: Start 1999-06; Primary Completion 2001-12 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
mobility score | 1 year
  questionnaire to nurses in charge of nursing home patients on specific items on mobility, which were used to create mobility score
socialization score | 1 year
  questionnaire to nurses in charge of nursing home patients on items specific to subject socialization, used to create socialization score

CONTACTS AND LOCATIONS:
Overall Officials: Sheila West, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman DS, Munoz B, Massof RW, Bandeen-Roche K, West SK. Grating visual acuity using the preferential-looking method in elderly nursing home residents. Invest Ophthalmol Vis Sci. 2002 Aug;43(8):2572-8. PMID 12147587
- [Background] West SK, Friedman D, Munoz B, Roche KB, Park W, Deremeik J, Massof R, Frick KD, Broman A, McGill W, Gilbert D, German P. A randomized trial of visual impairment interventions for nursing home residents: study design, baseline characteristics and visual loss. Ophthalmic Epidemiol. 2003 Jul;10(3):193-209. doi: 10.1076/opep.10.3.193.15081. PMID 12815493
- [Background] Friedman DS, West SK, Munoz B, Park W, Deremeik J, Massof R, Frick K, Broman A, McGill W, Gilbert D, German P. Racial variations in causes of vision loss in nursing homes: The Salisbury Eye Evaluation in Nursing Home Groups (SEEING) Study. Arch Ophthalmol. 2004 Jul;122(7):1019-24. doi: 10.1001/archopht.122.7.1019. PMID 15249367
- [Result] Friedman DS, Munoz B, Roche KB, Massof R, Broman A, West SK. Poor uptake of cataract surgery in nursing home residents: the Salisbury Eye Evaluation in Nursing Home Groups study. Arch Ophthalmol. 2005 Nov;123(11):1581-7. doi: 10.1001/archopht.123.11.1581. PMID 16286622